CLINICAL TRIAL: NCT02591784
Title: The Phase II of Nimotuzumab in Combination With Radiotherapy for Esophageal Cancer
Brief Title: Nimotuzumab in Combination With Radiotherapy for Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT-IST-ESO-002
Record Dates: First submitted 2015-08-17; First posted 2015-10-30 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2015-08

CONDITIONS: Esophageal
Keywords: nimotuzumab esophageal radiotherapy
MeSH Terms: interventions — nimotuzumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nimotuzumab group (Experimental): Nimotuzumab+radiotherapy
  Interventions: Drug: Nimotuzumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Nimotuzumab — the nimotuzumab treatment; 200mg/w,weekly,5-6 weeks.
Radiation: Radiotherapy — the Radiotherapy treatment;95%PTV A dose of 50-60Gy will be administered in 25-30 fractions ( 2 Gy /fraction)

SUMMARY:
Nimotuzumab (hR3) is an IgG1 humanized monoclonal antibody that recognized an epitope located in the extra cellular domain of the human epidermal growth factor receptor (EGFR). Clinical efficacy has been shown in adult with head and neck cancer. The phase II study assessed the efficacy and safety of the combination of Nimotuzumab administered concomitantly with radiotherapy in patients with esophageal cancer tumours.

DETAILED DESCRIPTION:
Clinical efficacy has been shown in adult with head and neck cancer. The phase II study assessed the efficacy and safety of the combination of Nimotuzumab administered concomitantly with radiotherapy in patients with esophageal cancer tumours.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically or cytology diagnosed phase II-III esophageal carcinoma or IV thoracic segments carcinoma with the supraclavicular lymph nodes metastasis.
2. with the measureable lesion of the newly diagnosed the esophageal carcinoma.
3. age 18-75 years old
4. ECOG≤2
5. Expect survival date ≥3 months
6. without serious diseases of important organs
7. signature in the inform consent.

Exclusion Criteria:

1. pregnant or breast-feeding women or using a prohibited contraceptive method.
2. with psychiatric diseases.
3. with serious diseases or uncontrolled infection.
4. with history of other tumors.
5. participation other clinical trials within 1 month prior to inclusion in the trial.
6. not the first antitumor treatment .

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The rate of AE(adverse event) or toxicity ( Both acute and chronic toxicity will be evaluated.) | 3 months
  assement of advers event after using medication based TAAE evaluation form

SECONDARY OUTCOMES:
Complete response | 3 months
Partial response (PR) | 3 months
Stable disease (SD) | 3 months
Progressive disease (PD) | 3 months
Median survival time (MST) | 2 years
Overall survival (OS) | 1 year,2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lvhua Wang, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (5):
- China (5):
  - The Affiliated tumour hosiptal of HARBIN Medical University, Harbin, Heilongjiang
  - Wuhan Union Hospital, Wuhan, Hubei
  - Qilu Hospital,Shandong University, Jinan, Shandong
  - Cancer Institute & Hospital, Chinese Academy of Medical Sciences, Beijing
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin